CLINICAL TRIAL: NCT06290102
Title: An Open Label, Single Dose, 3-Period, Crossover Study to Determine the Pharmacokinetic Profile and Safety of Fluticasone Propionate/Albuterol Sulfate (Fp/ABS) Multidose Dry Powder Inhaler With e-Module (eMDPI) Compared to Fluticasone Propionate Multidose Dry Powder Inhaler (Fp MDPI) in Participants With Asthma (4 to 11 Years Old)
Brief Title: Pharmacokinetic Profile and Safety of Fluticasone Propionate and Albuterol Sulfate in Combination When Compared to Fluticasone Propionate Multidose Dry Powder Inhaler (Fp MDPI) in Children Aged 4 to 11 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TV56248-RES-10204
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence ABC (Experimental)
  Interventions: Drug: TEV-56248; Drug: Fp MDPI
- Sequence BCA (Experimental)
  Interventions: Drug: TEV-56248; Drug: Fp MDPI
- Sequence CAB (Experimental)
  Interventions: Drug: TEV-56248; Drug: Fp MDPI
- Sequence ACB (Experimental)
  Interventions: Drug: TEV-56248; Drug: Fp MDPI
- Sequence BAC (Experimental)
  Interventions: Drug: TEV-56248; Drug: Fp MDPI
- Sequence CBA (Experimental)
  Interventions: Drug: TEV-56248; Drug: Fp MDPI

INTERVENTIONS:
Drug: TEV-56248 — Pharmaceutical form: Dry powder
  Route of administration: Oral inhalation
  Other Names: - fluticasone propionate/albuterol sulfate multidose dry powder inhaler with e-module (Fp/ABS eMDPI)
Drug: Fp MDPI — Pharmaceutical form: Dry powder
  Route of administration: Oral inhalation
  Other Names: - fluticasone propionate multidose dry powder inhaler

SUMMARY:
The primary objectives of this study are:

* To determine the pharmacokinetic (PK) profile of fluticasone propionate (Fp) and albuterol sulfate (ABS), delivered in combination, from a single dose of TEV-56248 (Fp and ABS multidose dry powder inhaler with e-module [Fp/ABS eMDPI]) in participants with asthma
* To compare the PK profiles of Fp for 2 different dose strengths of TEV-56248 to that of fluticasone propionate multidose dry powder inhaler (Fp MDPI)
* To compare the PK profiles of ABS between the 2 different strengths of TEV-56248

The secondary objective is:

• To evaluate the safety of a single dose of TEV-56248 and a single dose of Fp MDPI

DETAILED DESCRIPTION:
The planned duration for this trial is approximately 1.5 to 3 months. The trial includes a 14-day screening period, 3 treatment periods (2 days each), and a follow up visit 7 days after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of asthma as defined by the Global Initiative for Asthma guidelines (GINA 2023), which has been present for a minimum of 3 months and has been stable (defined as no exacerbations and no changes in asthma medication) for at least 30 days before the Screening Visit
* Has persistent asthma, with a forced expiratory value (FEV1) that is greater than or equal to 80% of the value predicted for age, height, sex, and race at the Screening Visit
* Demonstrate acceptable inhalation technique with the training inhaler
* Able to stop (as judged by the Investigator) his or her rescue medication, for approximately 6 hours before the Screening Visit and for approximately 4 hours before training sessions in periods 1-3
* Has body mass index (BMI) within the 3rd and 97th percentiles for the participant's age and gender. The participant must have a weight of ≥18 kilograms (kg)
* Able to achieve a peak inspiratory flow (PIF) rate of at least 60 liters per minute (L/min) on an inhaler training device

NOTE- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Participant has a history of a life-threatening asthma exacerbation that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest, or hypoxic seizures
* Has participated as a randomized participant in any investigational drug trial within 30 days (starting from the final follow-up visit of that trial) preceding the Screening Visit or plans to participate in another investigational drug trial at any time during this trial
* Known hypersensitivity to any corticosteroid, albuterol, or any of the ingredients in the investigational medicinal product
* Asthma exacerbation requiring systemic corticosteroids within 30 days of the Screening Visit, or has had any hospitalization for asthma within 2 months of the Screening Visit

NOTE- Additional criteria apply, please contact the investigator for more information

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Drug Concentration (Cmax) of Fluticasone Propionate (Fp) | Up to 24 hours postdose
Maximum Observed Plasma Drug Concentration (Cmax) of Albuterol Sulfate(ABS) | Up to 24 hours postdose
Area Under the Plasma Drug Concentration-Time Curve from Time 0 to the Time of the Last Measurable Drug Concentration (AUC0-t) for Fp | Up to 24 hours postdose
Area Under the Plasma Drug Concentration-Time Curve from Time 0 to the Time of the Last Measurable Drug Concentration (AUC0-t) for ABS | Up to 24 hours postdose
Area Under the Plasma Drug Concentration-Time Curve from Time 0 to 24 Hours Postdose (AUC0-24) of Fluticasone Propionate | Up to 24 hours postdose
AUC0-24 of Albuterol Sulfate | Up to 24 hours postdose
Time to Maximum Observed Plasma Drug Concentration (tmax) for Fp | Up to 24 hours postdose
Time to Maximum Observed Plasma Drug Concentration (tmax) for ABS | Up to 24 hours postdose
Terminal Phase (Apparent Elimination) Half-Life (t½) of Fp | Up to 24 hours postdose
Terminal Phase (Apparent Elimination) Half-Life (t½) of ABS | Up to 24 hours postdose
Last Measurable Concentration Above the Quantification Limit (Clast) of Fp | Up to 24 hours postdose
Last Measurable Concentration Above the Quantification Limit (Clast) of ABS | Up to 24 hours postdose
Time of Last Measurable Concentration (tlast) of Fp | Up to 24 hours postdose
Time of Last Measurable Concentration (tlast) of ABS | Up to 24 hours postdose

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 2 Months
Number of Participants with Serious Adverse Events (SAEs) | Up to 2 Months
Number of Participants Who Withdrawal From Trial Due to Treatment Emergent Adverse Events (TEAEs) | Up to 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (10):
- United States (10):
  - Teva Investigational Site 12010, Mobile, Alabama
  - Teva Investigational Site 12003, Long Beach, California
  - Teva Investigational Site 12007, Miami, Florida
  - Teva Investigational Site 12005, Miami, Florida
  - Teva Investigational Site 12002, Miami, Florida
  - Teva Investigational Site 12008, Lafayette, Louisiana
  - Teva Investigational Site 12011, Columbia, Missouri
  - Teva Investigational Site 12012, Oklahoma City, Oklahoma
  - Teva Investigational Site 12001, Boerne, Texas
  - Teva Investigational Site 12009, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.
URL: https://www.clinicalstudydatarequest.com/